CLINICAL TRIAL: NCT00004340
Title: Phase II Randomized Study of the Effects of Growth Hormone on Children and Adolescents on Maintenance Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Los Angeles (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11899; UCLA-612
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Renal Osteodystrophy; End Stage Renal Disease
Keywords: end stage renal disease; rare disease; renal and genitourinary disorders; renal osteodystrophy
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Kidney Failure, Chronic; Rare Diseases; Urogenital Diseases | interventions — Calcitriol; Growth Hormone

INTERVENTIONS:
Drug: calcitriol
Drug: growth hormone

SUMMARY:
OBJECTIVES: I. Evaluate the separate and combined skeletal effects of recombinant human growth hormone (GH) and calcitriol in patients with adynamic renal osteodystrophy.

II. Assess whether calcium-regulated changes in parathyroid hormone secretion predict changes in bone formation.

III. Characterize the response to GH in cancellous bone and in growth plate cartilage in patients with secondary hyperparathyroidism during calcitriol therapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by bone lesion turnover and secondary hyperparathyroidism.

Patients in the first group are treated with recombinant human growth hormone subcutaneously every day for 8 months.

Patients in the second group are treated with calcitriol for 8 months, administered as a daily oral dose or an intraperitoneal dose three times a week.

Patients in the third group are treated with growth hormone and calcitriol (same dosages as above).

A control group does not receive any hormonal therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* End-stage renal disease undergoing continuous cycling peritoneal dialysis at the University of California at Los Angeles

--Prior/Concurrent Therapy--

* No concurrent prednisone
* No concurrent cytotoxic agents
* At least 12 months since parathyroidectomy

--Patient Characteristics--

* Other: No documented history of poor compliance with medical treatment regimens

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Overall Officials: Isidro B. Salusky, Study Chair — University of California, Los Angeles
Locations (1):
- University of California Los Angeles School of Medicine, Los Angeles, California, United States